CLINICAL TRIAL: NCT01986946
Title: A Comparison of Epidural Analgesia With Standard Care Following Lumbar Spinal Fusion: A Prospective Randomized Study
Brief Title: Epidural Analgesia Versus IV Analgesia in Lumbar Spine Fusions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00041252
Record Dates: First submitted 2013-01-03; First posted 2013-11-19 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Lumbar Spine Fusion; Pain; Back Pain
MeSH Terms: conditions — Pain; Back Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous opioids (Experimental): This is the standard of care method for post-operative analgesia following lumbar spine fusion surgery. Participants randomly assigned to this arm will receive Intravenous Patient-Controlled Analgesia (IVPCA) with dilaudid (or other opioid) for post-operative pain control.
  Interventions: Drug: Dilaudid
- Epidural Catheter (Experimental): The intervention to be tested in this study against standard intravenous opioids is infusion of local anesthetic and dilaudid via epidural catheter for post-operative pain control in patients undergoing lumbar spine fusion surgery.
  Interventions: Other: Epidural Catheter - Dilaudid

INTERVENTIONS:
Other: Epidural Catheter - Dilaudid — Placement of an epidural catheter to administer local anesthetic and opioid (dilaudid) to the epidural space will be studied as compared to use of intravenous opioid (dilaudid) for pain control following lumbar spine fusion surgery.
  Arms: Epidural Catheter
Drug: Dilaudid — Patients in this arm will receive intravenous patient-controlled opioid analgesia (Dilaudid).
  Arms: Intravenous opioids

SUMMARY:
1. Protocol Title - A Comparison of Epidural Analgesia with Standard Care Following Lumbar Spinal Fusion: A Prospective Randomized Study
2. Purpose of the Study - This prospective randomized study will enroll 200 patients undergoing elective Lumbar Spinal Fusion at Duke University Hospital. The primary objective is to determine the effect of epidural analgesia, as compared with standard care, on post-operative analgesia.

Hypothesis:

The investigators hypothesize that patients undergoing Lumbar Spinal Fusion surgery with epidural catheter placement will have superior post-operative analgesia compared to patients undergoing standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are scheduled for elective Transforaminal Lumbar Interbody Fusion surgery

Exclusion Criteria:

* Baseline cognitive deficits sufficient to make objective pain self-assessments unreliable in the estimation of the Study Investigators.
* Inability to follow directions or comprehend the English language.
* Females who are pregnant as determined by positive pregnancy test on or before the day of surgery.
* Prisoners.
* Patient refusal to provide informed consent.
* Allergy to amide local anesthetics (lidocaine, bupivacaine, ropivacaine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Manning, MD/PhD, Principal Investigator — Duke University Hospital Department of Anesthesiology; Carlos Bagley, MD, Principal Investigator — Duke University Hospital Department of Neurosurgery
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Background] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Background] Abrishamkar S, Eshraghi N, Feizi A, Talakoub R, Rafiei A, Rahmani P. Analgesic effects of ketamine infusion on postoperative pain after fusion and instrumentation of the lumbar spine: a prospective randomized clinical trial. Med Arh. 2012;66(2):107-10. doi: 10.5455/medarh.2012.66.107-110. PMID 22486142
- [Background] Sekar C, Rajasekaran S, Kannan R, Reddy S, Shetty TA, Pithwa YK. Preemptive analgesia for postoperative pain relief in lumbosacral spine surgeries: a randomized controlled trial. Spine J. 2004 May-Jun;4(3):261-4. doi: 10.1016/j.spinee.2003.11.009. PMID 15125846
- [Background] Cohen BE, Hartman MB, Wade JT, Miller JS, Gilbert R, Chapman TM. Postoperative pain control after lumbar spine fusion. Patient-controlled analgesia versus continuous epidural analgesia. Spine (Phila Pa 1976). 1997 Aug 15;22(16):1892-6; discussion 1896-7. doi: 10.1097/00007632-199708150-00016. PMID 9280026
- [Background] Sucato DJ, Duey-Holtz A, Elerson E, Safavi F. Postoperative analgesia following surgical correction for adolescent idiopathic scoliosis: a comparison of continuous epidural analgesia and patient-controlled analgesia. Spine (Phila Pa 1976). 2005 Jan 15;30(2):211-7. doi: 10.1097/01.brs.0000150832.53604.64. PMID 15644759
- [Background] Yukawa Y, Kato F, Ito K, Terashima T, Horie Y. A prospective randomized study of preemptive analgesia for postoperative pain in the patients undergoing posterior lumbar interbody fusion: continuous subcutaneous morphine, continuous epidural morphine, and diclofenac sodium. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2357-61. doi: 10.1097/01.brs.0000184377.31427.fa. PMID 16261108
- [Background] Parker SL, Lerner J, McGirt MJ. Effect of minimally invasive technique on return to work and narcotic use following transforaminal lumbar inter-body fusion: a review. Prof Case Manag. 2012 Sep-Oct;17(5):229-35. doi: 10.1097/NCM.0b013e3182529c05. PMID 22850657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 participants consented in the study, 3 participants were not randomized in the study due to not having the surgery.
Period: Overall Study
Arm/Group | Intravenous Opioids | Epidural Catheter
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Opioids | Epidural Catheter | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 6 | 8
Gender [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain as Assessed by Visual Analogue Scale (VAS)
Description: The VAS scale ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain.
Time Frame: Postoperative day 1
Population: Participant that provided a VAS score at postoperative day 1 time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 3 | 8
units on a scale | 36.33 (26.66) | 40.63 (29.09)

2. Secondary Outcome: Patient Satisfaction With Perioperative Analgesia
Description: Patients will be assessed for satisfaction with their peri-operative analgesia in the recovery room and each day of their epidural infusion or intravenous opioid infusion by the Acute Pain Service, and at their surgical follow-up visit. Likert scale ranges from 1 to 5 (1=very satisfied and 5=Very Dissatisfied).
Time Frame: Post-operative Day 1
Population: Analyasis was completed on all participants who completed the patient satisfaction with perioperative analgesia assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 7
units on a scale | 2.4 (1.02) | 1.29 (0.7)

3. Secondary Outcome: Patient Satisfaction With Perioperative Analgesia
Description: as for outcome 2
Time Frame: 6-Week Follow up Visit
Population: Participants who completed the patient satisfaction scale at the 6 week follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 3 | 8
units on a scale | 2 (0.82) | 1.5 (0.71)

4. Secondary Outcome: Patient Satisfaction With Overall Care
Description: Likert scale ranges from 1 to 5 (1=very satisfied and 5=Very Dissatisfied).
Time Frame: 6-Week Follow up Visit
Population: Participants who completed the patient satisfaction scale at the 6 week follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 3 | 8
units on a scale | 1 (0) | 1.5 (0.71)

5. Secondary Outcome: Number of Participants With Events of Special Interest
Description: Patients will be assessed for development of a deep vein thrombosis after surgery, and surgical site infection.
Time Frame: Post-operative Day 30
Population: Data not collected
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events Related to the Study
Description: Patients will be assessed in the recovery room and each day of their epidural or intravenous opioid infusions, and at their surgical follow-up visit.
Time Frame: 6-week Follow up Visit
Measure: Number; unit: participants
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 9
participants | 0 | 0

7. Secondary Outcome: Total Post-operative Opioid Consumption
Time Frame: during hospitalization (approximately 3-8 days)
Measure: Mean (Standard Deviation); unit: oral morphine equivilant (mg)
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 9
oral morphine equivilant (mg) | 438.52 (292.87) | 410.42 (501.09)

8. Secondary Outcome: Number of Participants Experiencing Delirium
Time Frame: Post-operative Day 1
Population: Only participants who had assessment for delirium are include in the analysis.
Measure: Number; unit: participants
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 8
participants | 0 | 0

9. Secondary Outcome: Number of Participants Experiencing Delirium
Time Frame: Post-operative Day 2
Population: Participants who were evaluated for Delirium on Day 2
Measure: Number; unit: participants
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 6
participants | 0 | 0

10. Secondary Outcome: Number of Participants Experiencing Delirium
Time Frame: Post-operative Day 3
Population: Participants who were evaluated for Delirium on Day 3
Measure: Number; unit: participants
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 1 | 5
participants | 0 | 0

11. Secondary Outcome: Number of Participants Readmitted to Hospital Within 30 Days of Surgery
Time Frame: Post-operative Day 30
Measure: Number; unit: participants
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 9
participants | 0 | 0

12. Secondary Outcome: Length of Hospital Stay
Time Frame: during hospitalization (approximately 3-8 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 5 | 9
days | 4.4 (1.02) | 4.33 (1.41)

13. Secondary Outcome: Wound Infection Rates
Time Frame: during hospitalization (approximately 3-8 days)
Population: Data not collected
Arm/Group | Intravenous Opioids | Epidural Catheter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous Opioids | Epidural Catheter
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Opioids (N=5) | Epidural Catheter (N=9)
Hypotension (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment was terminated when co-PI/coordinator left Duke. No surgical collaborators would enroll subjects. Low enrollment of the study significantly affected the analysis, as both study arms were expected to have 100 participants each.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No